CLINICAL TRIAL: NCT05027828
Title: Circulating Tumor DNA as a Novel Molecular Marker of Treatment Efficacy to Guide Targeted Maintenance Therapy for Patients With High Grade Serous Ovarian Cancer
Brief Title: CtDNA as a Novel Biomarker of Treatment Efficacy in Patients With Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-21-008
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: High-grade Serous Ovarian Cancer; Circulating Tumor DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and whole blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients using olaparib only
- patients using olaparib combined with bevacizumab

SUMMARY:
This study is a prospective observational clinical trial. Patients who were diagnosed and treated for the first time were enrolled and their surgical pathology was confirmed to be high-grade serous ovarian cancer. At the same time, these patients will receive first-line maintenance treatment with PARP inhibitors after traditional chemotherapy. During the trial period, patients' plasma will be collected before surgery, after chemotherapy, during targeted maintenance therapy, and during disease progression, and ctDNA-specific genomes will be detected, and clinical data will be collected over the same period. It is expected that specific ctDNA can be used to predict the efficacy of PARP inhibitors in patients with ovarian cancer, and to detect the recurrence of the disease early.

ELIGIBILITY:
Inclusion Criteria:

1. Ovarian cancer first diagnosed and treated;
2. Pathologically confirmed as epithelial ovarian cancer/fallopian tube cancer/primary peritoneal cancer;
3. The stage of the disease is II-IV, and surgery will be performed after evaluation;
4. Age ≥ 18 years old;
5. Subjects and their families fully understand the research plan and sign an informed consent form.

Exclusion Criteria:

1. Pathologically confirmed as non-epithelial ovarian cancer;
2. Surgical treatment cannot be performed after evaluation;
3. Malignant tumors found in other parts of the study were found within five years before enrollment or at the time of enrollment;
4. Patients who do not agree to use clinical first-line targeted drugs;
5. Severe mental illness;
6. Severe cardiovascular disease, uncontrollable infection, or other uncontrollable comorbid diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly-diagnosed and treated patients with high-grade serous ovarian cancer who will receive PARP inhibitors as first-line maintenance therapy after surgery and traditional chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | about 36 months after using PARP inhibitors
  To determine the different prognosis of patients after using the PARP inhibitor for first-line maintenance treatment, at the same time, the plasma will be collected and tested for ctDNA before using the PARP inhibitor, during use and when the disease is progressing.

SECONDARY OUTCOMES:
Overall survival | about over 5 years after using PARP inhibitors
Objective response rate | 36 months after using PARP inhibitors
  To evaluate the general response of patients with ovarian cancer to PARP inhibitors

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China